CLINICAL TRIAL: NCT00563121
Title: Vascular Endothelial Growth Factor Levels in Aqueous, Vitreous and Subretinal Fluid in Patients With Retinopathy of Prematurity Stage IV and V
Brief Title: VEGF Levels in Aqueous, Vitreous and Subretinal Fluid in ROP Stage IV and V
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ROP001
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Retinopathy of Prematurity
Keywords: Retinopathy of Prematurity; ROP; Vascular Endothelial Growth Factor; VEGF; Vitreous; Subretinal Fluid; ELISA; VEGF levels in Aqueous, Vitreous and subretinal Fluid
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Vitrectomy — Open-Sky vitrectomy, with resection of the tunica vasculosa lentis, and retinal reattachment

SUMMARY:
To determine the degree of VEGF in Aqueous, vitreous and SRF in patients with ROP in stage V. Verifying that it is greater to that found in healthy newborn patients with different ocular pathology.

DETAILED DESCRIPTION:
Introduction:

Vascular Endothelial Growth Factor (VEGF) is a dimeric glycoprotein, naturally expressed in epithelial and tumor cells (1). In conditions of hypoxia it is secreted by the pericytes, the Retina Pigmented epithelium (RPE)and glial cells, including a the Müller cells (1,2,4,5) favoring the formation of new abnormal vessels (1). Its activity is mediated by two high affinity receptors: the receptor VEGF 1 (FLT-1) and VEGF 2 (FLT-2) (1,9). The FLT-1 promotes cellular proliferation whereas FLT-2 the migration and cell- extracellular matrix interaction (9). The VEGF is essential as much for the normal retinal vascularization as for pathological (5,14).

Normal Retinal vascularization has two phases: In the first fase, cells of mesenquimatous origin form the first superficial plexus (14-21 weeks of gestation). In the second phase, denominated "angiogenesis phase", the superficial and deep capillary plexus are formed (15,20). The second phase is highly dependent of VEGF induced by hypoxia (15,20). In the normal retina the growth occurs from the optical nerve to the periphery (17).

The scientific progress in the neonatal intensive care units in the last years has allowed the survival of a larger number of premature newborns(15).

The Retinopathy of Prematurity (ROP)(ROP) was described for the first time in 1942 (4), at the present moment it is a public health problem in the developing countries. Of each 100.000 blind child in Latin America, 24.000 are due to ROP (240/1000 blind child) (17). It is the main cause of blindness in premature new born (1,4,5). It is of multifactorial etiology (17) but it has been related to a short gestational age (smaller to 32 weeks of gestation) (4), to low birth weight (less of 1500gr) or very low birth weight (less 1250gr)(1,4,5,17,18,20), to the administration of high oxygen concentration immediately after birth (1,3,18), low levels of the Insulin-like growth factor(IGF-I) and excessive production of VEGF (3,17).

All this, combined with large periods of hyperoxia-hypoxia, Produces that the normal vascularization of the retina stops. This also produces vascular-occlusive changes, arteriovenous anastomoses in the edge of the vascularized with the none-vascularized retina (18), begins the formation of abnormal vessels towards the vitreous, finally lead to retina detachment in the most severe cases (2,3,4,5).

The International Classification of ROP classifies it in 5 stages, dividing it in 3 anatomical zones. A threshold stage is considered when we have the presence of stage 3, in zone 1 or 2 in 5 continuous hour uses or 8 discontinuous with plus disease (15,16,17). The pre-threshold stage is divided in two types: type 1 is any stage of the disease in zone 1 with plus disease, stage 3, without plus disease in zone 1 or stage 2 or 3 with plus in zone 2. Type 2 is stage 1 or 2 without plus disease in zone 1 or stage 3 without plus disease in zone 2 (17,19). The threshold stage happens approximately in 5% of the patients with very low weight to the birth, of which the 10-15% develop blindness (6,8)

It is a public health problem that continuous without having an effective prophylaxis (5), nevertheless the use of constant oxygen concentrations, avoiding the periods of hyperoxia-hypoxia, has demonstrated to produce a decrease of the presentation of advanced stages of the disease and the necessity of ophthalmological surgery (5). The early diagnosis and treatment in thresholds stages have changed the prognosis of this disease (11,12). The use of the laser as treatment in the threshold and prethreshold stages is successful in the 91-95% of the cases(10), the ablative effect on the neurons, probably diminishes the VEGF production (15). The use of the vitrectomy in the early cases of retinal detachment also has good results (13).

For the determination and the quantification of VEGF several laboratory techniques have been used, as they are the Westernblot (1), the flow cytometry (7), CBA (7). Nevertheless, the Enzyme-linked immunoabsorbent assay (ELISA) remains the gold standard for the measurement of interleukins, growth factors and other cytokines in corporal fluids, including the vitreous, Aqueous and subretinal fluid (1,5,7).

It has been demonstrated in humans that there are high vitreous concentrations of VEGF in eyes with active neovascularization (6,14). In the same way, the animal models of ROP report high levels of VEGF (2,21). The levels of this growth factor are altered in both stages, with a more marked increase during the first stage (2). Some clinical studies in patients with ROP in stage 4 and 5 have reported an increase of up to 90 times greater of the concentration of VEGF in the subretinal liquid in comparison with the found in patients with retinal detachment of any other cause (1). Finally, when it has been possible to examine retinas immediately after the treatment (due to death of the patient) have been found a low expression of mRNA of VEGF in the treated cells (6).

Problem:

In spite of the great amount of animals models and some clinical tests in humans. Until now there are no data in the world-wide Literature that report, in a specific way, the VEGF concentrations in the different compartments of the eye, during the active stage of the ROP. Also a comparison between the concentration of this growth factor found in the ROP patients with, the level found in other well characterized pathologies that also produce VEGF, as it is Diabetes Mellitus (DM) does not exist

ELIGIBILITY:
Inclusion Criteria:

* Premature newborns with less than 32 weeks of gestation.
* Low birth weight (less than 1500gr)
* Stage V ROP.
* The parents has signed the informed consent.

Exclusion Criteria:

* Previous treatment of ROP.
* Surgery or another ocular pathology of any type.
* Systemic diseases, including diabetes mellitus, congestive heart failure acute renal insufficiency, Chronic renal insufficiency, high blood pressure.
* Lack of Informed consent.

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2007-03 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
VEGF Levels | one day

CONTACTS AND LOCATIONS:
Overall Officials: Raul Velez-Montoya, MD, Principal Investigator — Asociación para Evitar la Ceguera en Mexico; Hugo Quiroz-Mercado, MD, Principal Investigator — Asociación para Evitar la Ceguera en Mexico
Locations (2):
- Mexico (2):
  - Asociación para Evitar la Ceguera en Mexico, Mexico City, Mexico City
  - Asociacion Para Evitar la Ceguera en Mexico. Hospital Luis Sanchez Bulnes, Mexico City, Mexico D. F.

REFERENCES:
- [Background] Lashkari K, Hirose T, Yazdany J, McMeel JW, Kazlauskas A, Rahimi N. Vascular endothelial growth factor and hepatocyte growth factor levels are differentially elevated in patients with advanced retinopathy of prematurity. Am J Pathol. 2000 Apr;156(4):1337-44. doi: 10.1016/S0002-9440(10)65004-3. PMID 10751359
- [Background] Pierce EA, Foley ED, Smith LE. Regulation of vascular endothelial growth factor by oxygen in a model of retinopathy of prematurity. Arch Ophthalmol. 1996 Oct;114(10):1219-28. doi: 10.1001/archopht.1996.01100140419009. PMID 8859081
- [Background] Gaynon MW. Rethinking STOP-ROP: is it worthwhile trying to modulate excessive VEGF levels in prethreshold ROP eyes by systemic intervention? A review of the role of oxygen, light adaptation state, and anemia in prethreshold ROP. Retina. 2006 Sep;26(7 Suppl):S18-23. doi: 10.1097/01.iae.0000244292.86627.1e. PMID 16946672
- [Background] Hellstrom A, Perruzzi C, Ju M, Engstrom E, Hard AL, Liu JL, Albertsson-Wikland K, Carlsson B, Niklasson A, Sjodell L, LeRoith D, Senger DR, Smith LE. Low IGF-I suppresses VEGF-survival signaling in retinal endothelial cells: direct correlation with clinical retinopathy of prematurity. Proc Natl Acad Sci U S A. 2001 May 8;98(10):5804-8. doi: 10.1073/pnas.101113998. Epub 2001 May 1. PMID 11331770
- [Background] Modanlou HD, Gharraee Z, Hasan J, Waltzman J, Nageotte S, Beharry KD. Ontogeny of VEGF, IGF-I, and GH in neonatal rat serum, vitreous fluid, and retina from birth to weaning. Invest Ophthalmol Vis Sci. 2006 Feb;47(2):738-44. doi: 10.1167/iovs.05-1046. PMID 16431975
- [Background] Cooke RW, Drury JA, Mountford R, Clark D. Genetic polymorphisms and retinopathy of prematurity. Invest Ophthalmol Vis Sci. 2004 Jun;45(6):1712-5. doi: 10.1167/iovs.03-1303. PMID 15161830
- [Background] Maier R, Weger M, Haller-Schober EM, El-Shabrawi Y, Theisl A, Barth A, Aigner R, Haas A. Application of multiplex cytometric bead array technology for the measurement of angiogenic factors in the vitreous. Mol Vis. 2006 Oct 2;12:1143-7. PMID 17093399
- [Background] Phelps DL; ETROP Cooperative Group. The Early Treatment for Retinopathy of Prematurity study: better outcomes, changing strategy. Pediatrics. 2004 Aug;114(2):490-1. doi: 10.1542/peds.114.2.490. No abstract available. PMID 15286235
- [Background] Yoo MH, Hyun HJ, Koh JY, Yoon YH. Riluzole inhibits VEGF-induced endothelial cell proliferation in vitro and hyperoxia-induced abnormal vessel formation in vivo. Invest Ophthalmol Vis Sci. 2005 Dec;46(12):4780-7. doi: 10.1167/iovs.05-0376. PMID 16303979
- [Background] Multicenter trial of cryotherapy for retinopathy of prematurity. Preliminary results. Cryotherapy for Retinopathy of Prematurity Cooperative Group. Arch Ophthalmol. 1988 Apr;106(4):471-9. doi: 10.1001/archopht.1988.01060130517027. PMID 2895630
- [Background] Itakura H, Kishi S, Kotajima N, Murakami M. Persistent secretion of vascular endothelial growth factor into the vitreous cavity in proliferative diabetic retinopathy after vitrectomy. Ophthalmology. 2004 Oct;111(10):1880-4. doi: 10.1016/j.ophtha.2004.03.035. PMID 15465550